CLINICAL TRIAL: NCT05281588
Title: Effects of Micro-osteoperforations on the Upper Incisors' Retraction: a Randomized Clinical Trial
Brief Title: Evaluation of Micro-osteoperforations to Accelerate Orthodontic Tooth Movement
Acronym: MOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontifícia Universidade Católica de Minas Gerais (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Micro-osteoperforations
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Orthodontic Tooth Movement
Keywords: Micro-osteoperforations; Orthodontic incisors retraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micro-osteoperforations (Experimental): Micro-osteoperforations- assisted upper incisors retraction
  Interventions: Procedure: Micro-osteoperforations
- Control (No Intervention): Upper incisors retraction not associated with any clinical intervention to accelerate tooth movement

INTERVENTIONS:
Procedure: Micro-osteoperforations — All micro-osteoperforations were performed only one time in the experimental group on the same day of the installation of the upper incisors' retraction mechanics. Perforations were performed with an individualized surgical guide and a 1.6 mm diameter stainless steel surgical drill perpendicular to the alveolar bone, 3 mm deep on the buccal surface, and 5 mm, on the palate. The depth of the perforations was controlled and standardized by a cursor developed and patented by the research group. Two micro-osteoperforations were aligned vertically distally from each upper incisor. Due to the proximity of the roots in the cervical third, only the most apical perforation was performed between the two central incisors. The first perforation was performed 6 mm away from the gingival margin, and the second, 5 mm from the first, in the vertical direction.
  Other Names: MOP
  Arms: Micro-osteoperforations

SUMMARY:
This clinical trial evaluated the efficacy of micro osteoperforations in accelerating the retraction of maxillary incisors.

DETAILED DESCRIPTION:
This single-centered randomized clinical trial evaluated the effects of micro-osteoperforations in the retraction of maxillary incisors in patients who required the extraction of the first premolars to correct malocclusion. The canine retraction was performed in a previous step. The possible effects of micro-osteoperforantions in the following parameters were evaluated in the upper arch: anteroposterior incisors and first molars displacement, space closure, inclination and length of central incisors.

ELIGIBILITY:
Inclusion Criteria:

* both male and female subjects
* 16 or more years old
* orthodontic need of upper incisors extractions
* presence of all upper permanent teeth with exception of the third molars.

Exclusion Criteria:

* diseases and medications that were likely to affect bone biology
* pregnancy
* poor oral hygiene
* previous orthodontic treatment
* evidence of bone loss
* active periodontal disease
* smoking
* syndromes or cleft patients
* severe crowding or Class II malocclusion (Pg-Nper > 18 mm, ANB > 7º, SN-GoGn > 38º e overjet > 10 mm).

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Anteroposterior displacement of the upper incisors | Up to 4 months
  The anteroposterior displacement of the upper incisors was assessed on superimposed digital models through the distance of points on the incisal edge and palatal cervical margin of these teeth to a coronal reference plan created on the initial CBCT scan.
Space closure | Up to 4 months
  The space closure was assessed by the distance between the most menial point of the medial surface of the canine to the most distal point of the distal surface of the lateral incisor.

SECONDARY OUTCOMES:
First molars anchorage loss | Up to 4 months
  The first molars anchorage loss was assessed on superimposed digital models through the distance of a point on the mesiobuccal cuspid to a coronal reference plan created on the initial CBCT scan.
Changes of the inclination of the central incisors | Up to 4 months
  The initial and final CBCT were superimposed by the "voxel-based method" in the Dolphin Imaging software (Chatsworth, CA, USA), using the cranial base as reference. The inclination of the central incisors was then assessed by means of the angle formed by the long axis of each central incisor in the initial and final CBCT.
Changes of the length of the central incisors | Up to 4 months
  The initial and final length of the central incisors were measured by creating a 2D line, passing through the lowest point of the incisal edge and the highest point of the root apex. To perform these measurements, a sagittal cut was used in which the longest length of these teeth was seen.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo V Soares, PhD, Study Director — Pontifícia Universidade Católica de Minas Gerais
Locations (1):
- Pontifícia Universidade Católica de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The research can be shared with others researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year
Access Criteria: All researchers

REFERENCES:
- [Derived] Mordente CM, Dores LS, Oliveira DD, Palomo JM, Souki BQ, Soares RV. Third Palatal Rugae as Stable Landmarks for Intraoral Models' Superimposition in Extraction Cases: A Retrospective Cohort Study. Orthod Craniofac Res. 2025 Dec 25. doi: 10.1111/ocr.70078. Online ahead of print. PMID 41445469